CLINICAL TRIAL: NCT03732963
Title: Oral Melatonin as Premedication During Monitored Anaesthesia Care for Patients Undergoing Loco-regional Chronic Subdural Hematoma Evacuation, a Randomized Controlled Trial
Brief Title: Oral Melatonin as Premedication During MAC for Patients Undergoing Loco-regional Chronic Subdural Hematoma Evacuation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N 45-2018/Ms
Record Dates: First submitted 2018-09-04; First posted 2018-11-07 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Monitored Anaesthesia Care; Loco-regional Chronic Subdural Hematoma Evacuation
Keywords: Oral Melatonin Premedication
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: (N-acetyl-5-methoxytryptamine) is a neurohormone secreted by the pineal gland. It is primarily responsible for the sleep awake cycle as its level decreases in the morning and increases by night; owing to reduced light intensity, leading to circadian rhythm. It provides circadian and seasonal timing through activation of G protein-coupled receptors (GPCRs) in target tissues. Melatonin exerts its hypnotic effects through the activation of the MT1 and MT2 melatonin receptors
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be done via computer generated numbers and concealed by serially numbered, opaque and sealed envelopes. The details of series will be unknown to the investigators and the group assignment will be kept in a set of concealed envelopes each bearing only the case number on the outside. Prior to the start of the study, the appropriately numbered envelopes will be opened by the nurse, the card will determine the assigned intervention for each patient, which will be prepared by a clinical pharmacist with no other role in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Group P) (Placebo Comparator): Group P: 20 patients will receive a placebo tablet preoperatively.
  Interventions: Drug: Placebo (Group P)
- Melatonin (Group M) (Active Comparator): Group M: 20 patients will receive an oral melatonin tablet 10 mg preoperatively.
  Interventions: Drug: Melatonin (Group M)

INTERVENTIONS:
Drug: Placebo (Group P) — Group P: 20 patients will receive a placebo tablet preoperatively.
  Other Names: Placebo Group
  Arms: Placebo (Group P)
Drug: Melatonin (Group M) — Group M: 20 patients will receive an oral melatonin tablet 10 mg preoperatively.
  Other Names: Melatonin Group
  Arms: Melatonin (Group M)

SUMMARY:
investigators assume that administration of preoperative melatonin will reduce the required dose of propofol in participants undergoing loco-regional chronic subdural hematoma evacuation, it may as well provide better postoperative analgesia and decrease the incidence of delirium.

DETAILED DESCRIPTION:
A number of studies showed that premedication with melatonin was associated with sedation without impairment of cognitive and psychomotor skills or prolonging recovery. Some studies demonstrated that melatonin decreases the amount of propofol required to produce an adequate depth of hypnosis at induction time

The effects of the oral administration of melatonin on the dose of propofol sedation in participants undergoing loco-regional chronic subdural hematoma evacuation have not been documented before.

The present study will be conducted to detect the efficacy of oral administration of melatonin on the reduction of the sedative dose of propofol in participants undergoing loco-regional chronic subdural hematoma evacuation.

ELIGIBILITY:
Inclusion Criteria:

* 50 -65 years
* ASA grade I to II
* Both sexes
* Patients with unilateral chronic subdural hematoma
* Patients who are vitally stable
* Glascow coma scale 14-15

Exclusion Criteria:

* Age below 50 and above 65 years.
* Gastro intestinal tract impractabililty.
* Patients with any substance abuse.
* Patients with hepatic or renal insufficiency.
* Patients on antipsychotic, anticonvulsant or anti-parkinsonian medication.
* Vitally unstable patients who cannot tolerate propofol sedation.
* Patients with known allergies to any of the drugs used.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
To compare propofol consumption among both groups. | 24 hours Postoperative
  propofol consumption per mg among both groups.

SECONDARY OUTCOMES:
Vital Signs | 24 hours Postoperative
  Blood pressure (mmHg) .
Number of intraoperative patients movements. | 24 hours Postoperative
  Intraoperative patients movements
Anesthesia recovery times /Hour in both groups. | 24 hours Postoperative
  Anesthesia recovery times in both groups
VAS score for pain in each group | 24 hours Postoperative
  VAS score for pain in each group
Time to first rescue analgesic in both groups. | 24 hours Postoperative
  Time to first rescue analgesic in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not Now